CLINICAL TRIAL: NCT02019550
Title: A Phase IV, Randomized, Prospective, US-based, Multicenter, Cross-over Study Evaluating Subject Ease-of-use With Rebif® Rebidose® and Rebiject II® Autoinjectors in Subjects With Relapsing Remitting Multiple Sclerosis (RRMS) Treated With REBIF® 44 mcg Subcutaneously Three Times a Week
Brief Title: Rebif® Rebidose® Versus Rebiject II® Ease-of-Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200136-573
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Rebif®Rebidose®; Rebiject II®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Rebif Rebidose, Then Rebiject II (Experimental): Subjects will self-inject Rebif at a dose of 44 microgram (mcg) subcutaneously three times a week by using Rebif Rebidose self-injector device in Treatment Period 1 for 4 weeks followed by self-injecting Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in Treatment Period 2 (4 weeks) for the next 4 weeks.
  Interventions: Device: Rebif Rebidose; Device: Rebiject II
- First Rebiject II, Then Rebif Rebidose (Experimental): Subjects will self-inject Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in Treatment Period 1 for 4 weeks followed by self-injecting Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebif Rebidose self-injector device in Treatment Period 2 for the next 4 weeks.
  Interventions: Device: Rebif Rebidose; Device: Rebiject II

INTERVENTIONS:
Device: Rebif Rebidose — Rebif 44 mcg will be injected subcutaneously three times a week using Rebif Rebidose self-injector device.
Device: Rebiject II — Rebif 44 mcg will be injected subcutaneously three times a week using Rebiject II self-injector device.

SUMMARY:
This is a Phase 4, prospective, open-label, randomized, cross-over, multicenter trial to evaluate ease-of-use with Rebif® Rebidose® and Rebiject II® autoinjectors in subjects with relapsing remitting multiple sclerosis (RRMS). Subjects will participate in the study for up to 10 weeks (including screening and treatment periods). The treatment period will last 8 weeks and include 12 self-injections using the Rebif® Rebidose® device and 12 self-injections using the Rebiject II® device.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 to 65 years of age inclusive, at the time of informed consent signature
* Diagnosis of RRMS
* Receiving Rebif®, 44 microgram subcutaneously three times a week, by manual injection for at least 12 weeks before the screening assessment and previous use of either Rebif® Rebidose® or Rebiject II® devices is acceptable if they have not been using them for the past 12 weeks prior to study entry and if, in the judgment of the investigator, the subjects are not experienced users
* Subject is capable of self-injecting using Rebif® Rebidose® and Rebiject II® injection devices
* Subject is willing and able to comply with the study procedures for the duration of the trial
* Signed, informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization before any trial-related activities are performed
* Female subjects of childbearing potential must have a negative pregnancy test at screening to be included in the trial and must be willing to avoid pregnancy by using a highly effective method of contraception
* Outpatient status at the time of screening
* Stable disease status without a history of surgical procedure or hospitalization within 30 days prior to Study Day 1, and with no surgical intervention planned for the duration of the study

Exclusion Criteria:

* Received MS therapy other than Rebif® within the 12 weeks before screening or at any time during the trial
* Inadequate liver function and bone marrow reserve as defined in the protocol
* Current complete transverse myelitis, bilateral optic neuritis, or neuromyelitis optica
* History of injection-site necrosis within 12 months before study entry
* History of alcohol or drug abuse in the past year
* Any autoimmune disorder, except for thyroid disease stable on medication
* Subject having moderate to severe renal impairment, in the Investigator's opinion.
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS
* Participation in another clinical trial within the past 30 days or an interventional trial for MS in the past 12 weeks
* Use of high-dose steroids within 14 days of screening
* Currently experiencing moderate to severe active inflammatory skin disease at sites of expected Rebif® injections
* History of clinically significant lipoatrophy at sites of expected Rebif® injections, in the investigator's opinion
* Current major depression or suicidal ideation or suicide attempt in the past year
* Experiencing spasticity which in the opinion of the Investigator, could interfere with self-injections
* Pregnant or lactating
* Inability to self-inject or visual impairment which, in the opinion of the Investigator, is severe enough, even with correction, to impede the subject's participation in this study
* Upper extremity deficit which, in the opinion of the Investigator, is severe enough to impede the subject's participation in this study
* Cognitive deficit which, in the opinion of the Investigator, is severe enough to impede the subject's participation in this study
* Subject-reported reason that he/she cannot complete the 8-week study
* Any other medical condition, which in the opinion of the Investigator makes the subject unsuitable for this study
* Known hypersensitivity to the trial treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (21):
- United States (21):
  - Research site, Cullman, Alabama
  - Research Site, Tuscon, Arizona
  - Research Site, Newport Beach, California
  - Research site, Fort Collins, Colorado
  - Research Site, Dover, Delaware
  - Research Site, Miami, Florida
  - Research site, Sunrise, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research site, Foxborough, Massachusetts
  - Research site, Golden Valley, Minnesota
  - Research Site, Stratford, New Jersey
  - Research Site, Patchogue, New York
  - Research Site, Hickory, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Greensburg, Pennsylvania
  - Research site, Spartanburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research site, Mansfield, Texas

REFERENCES:
- [Derived] Wray S, Hayward B, Dangond F, Singer B. Ease of use of two autoinjectors in patients with multiple sclerosis treated with interferon beta-1a subcutaneously three times weekly: results of the randomized, crossover REDEFINE study. Expert Opin Drug Deliv. 2018 Feb;15(2):127-135. doi: 10.1080/17425247.2018.1407755. Epub 2017 Dec 5. PMID 29206056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 sites in the United States.
Pre-assignment Details: Overall, 103 subjects were screened, for inclusion in this trial. Of which, 97 subjects were randomized into the study.
Groups:
- First Rebif Rebidose, Then Rebiject II: Subjects self-injected Rebif at a dose of 44 microgram (mcg) subcutaneously three times a week by using Rebif Rebidose self-injector device in Treatment Period 1 for 4 weeks followed by self-injecting Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in Treatment Period 2 for the next 4 weeks.
- First Rebiject II, Then Rebif Rebidose: Subjects self-injected Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in Treatment Period 1 for 4 weeks followed by self-injecting Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebif Rebidose self-injector device in Treatment Period 2 for the next 4 weeks.
Period: Treatment Period 1 (4 Weeks)
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Started | 46 | 51
Completed | 46 | 50
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 2 (4 Weeks)
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Started | 46 | 50
Completed | 46 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment.
Groups:
- First Rebif Rebidose, Then Rebiject II: Subjects self-injected Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebif Rebidose self-injector device in Treatment Period 1 for 4 weeks followed by self-injecting Rebif at a dose of 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in Treatment Period 2 for the next 4 weeks.
- Total: Total of all reporting groups
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose | Total
Number analyzed (Participants) | 46 | 51 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (9.78) | 47.5 (11.20) | 48.4 (10.54)
Gender [Count of Participants; unit: Participants]
  Female | 40 | 32 | 72
  Male | 6 | 19 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Rating Each Device as "Easy/Very Easy to Use" Based on User Trial Questionnaire (UTQ) at Week 4
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their overall experience with using the device as "very difficult", "difficult", "neither easy nor difficult", "easy", or "very easy". Percentage of subjects who rated the overall use of device as "easy" or "very easy" were reported. Here results are presented by device sequence.
Time Frame: Week 4
Population: FAS included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Easy | 34.8 | 50.0
  Very easy | 39.1 | 30.0

2. Primary Outcome: Percentage of Subjects Rating Each Device as "Easy/Very Easy to Use" Based on User Trial Questionnaire (UTQ) at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Easy | 45.7 | 24.0
  Very easy | 30.4 | 40.0

3. Primary Outcome: Percentage of Subjects Rating Each Device as "Easy/Very Easy to Use" Based on User Trial Questionnaire (UTQ) up to Week 8
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their overall experience with using the device as "very difficult", "difficult", "neither easy nor difficult", "easy", or "very easy". Percentage of subjects who rated the overall use of device as "easy" or "very easy" were reported. Here results are presented by device used.
Time Frame: Baseline up to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Rebif Rebidose: Subjects who were injected with Rebif 44 mcg subcutaneously three times a week by using Rebif Rebidose self-injector device in either Treatment Period 1 or 2.
- Rebiject II: Subjects who were injected with Rebif 44 mcg subcutaneously three times a week by using Rebiject II self-injector device in either Treatment Period 1 or 2.
Arm/Group | Rebif Rebidose | Rebiject II
Number analyzed (Participants) | 96 | 96
percentage of subjects
  Easy | 29.2 | 47.9
  Very easy | 39.6 | 30.2

4. Secondary Outcome: Number of Subjects Rating Each Device on Level of Satisfaction With Using the Device While Traveling Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of satisfaction with using the device while traveling (defined as being away from home overnight). Subjects assessed if they were satisfied with their ability to use the device while traveling overnight as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: FAS included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment. Here "Number of Participants Analyzed" = subjects evaluable for this outcome, "Number Analyzed"=subjects evaluable at the specified time point.
Measure: Number; unit: subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 17 | 21
subjects
  Week 4: Strongly disagree: number analyzed (Participants) | 17 | 18
  Week 4: Strongly disagree | 0 | 0
  Week 4: Disagree: number analyzed (Participants) | 17 | 18
  Week 4: Disagree | 0 | 0
  Week 4: Neither agree nor disagree: number analyzed (Participants) | 17 | 18
  Week 4: Neither agree nor disagree | 2 | 1
  Week 4: Agree: number analyzed (Participants) | 17 | 18
  Week 4: Agree | 5 | 7
  Week 4: Strongly agree: number analyzed (Participants) | 17 | 18
  Week 4: Strongly agree | 10 | 10
  Week 8: Strongly disagree: number analyzed (Participants) | 16 | 21
  Week 8: Strongly disagree | 1 | 0
  Week 8: Disagree: number analyzed (Participants) | 16 | 21
  Week 8: Disagree | 0 | 0
  Week 8: Neither agree nor disagree: number analyzed (Participants) | 16 | 21
  Week 8: Neither agree nor disagree | 1 | 3
  Week 8: Agree: number analyzed (Participants) | 16 | 21
  Week 8: Agree | 8 | 9
  Week 8: Strongly agree: number analyzed (Participants) | 16 | 21
  Week 8: Strongly agree | 6 | 9

5. Secondary Outcome: Percentage of Subjects Rating Each Device on Amount of Time Needed to Complete the Injection Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of satisfaction with respect to the amount of time it took to complete injection with the device. Subjects assessed if they were satisfied as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: FAS included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment. Here "Number of Participants Analyzed" signifies subjects evaluable for this outcome.
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 0.0 | 0.0
  Week 4: Disagree | 2.2 | 8.0
  Week 4: Neither agree nor disagree | 10.9 | 8.0
  Week 4: Agree | 39.1 | 50.0
  Week 4: Strongly agree | 47.8 | 34.0
  Week 8: Strongly disagree | 2.2 | 4.0
  Week 8: Disagree | 6.5 | 2.0
  Week 8: Neither agree nor disagree | 0.0 | 4.0
  Week 8: Agree | 50.0 | 44.0
  Week 8: Strongly agree | 41.3 | 46.0

6. Secondary Outcome: Percentage of Subjects Rating Each Device on Number of Steps Involved in Completing the Injection Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of satisfaction with respect to number of steps it took to complete an injection with the device. Subjects assessed if they were satisfied as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 0.0 | 2.0
  Week 4: Disagree | 0.0 | 10.0
  Week 4: Neither agree nor disagree | 0.0 | 20.0
  Week 4: Agree | 52.2 | 42.0
  Week 4: Strongly agree | 47.8 | 26.0
  Week 8: Strongly disagree | 2.2 | 4.0
  Week 8: Disagree | 6.5 | 4.0
  Week 8: Neither agree nor disagree | 8.7 | 4.0
  Week 8: Agree | 45.7 | 38.0
  Week 8: Strongly agree | 37.0 | 50.0

7. Secondary Outcome: Percentage of Subjects Rating Each Device on Ease of Holding Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their overall experience with holding the device as "very difficult", "difficult", "neither easy nor difficult", "easy", or "very easy". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: very difficult | 0.0 | 0.0
  Week 4: difficult | 4.3 | 6.0
  Week 4: neither easy nor difficult | 21.7 | 18.0
  Week 4: easy | 43.5 | 48.0
  Week 4: very easy | 30.4 | 28.0
  Week 8: very difficult | 0.0 | 4.0
  Week 8: difficult | 6.5 | 12.0
  Week 8: neither easy nor difficult | 13.0 | 20.0
  Week 8: easy | 43.5 | 28.0
  Week 8: very easy | 37.0 | 36.0

8. Secondary Outcome: Number of Subjects Rating Each Device on Level of Satisfaction With Using the Device Away From Home Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of satisfaction with using the device while away from home. Subjects assessed if they were satisfied with their ability to use the device while away from home as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 4
Measure: Number; unit: subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 17 | 18
subjects
  Week 4: Strongly disagree: number analyzed (Participants) | 11 | 18
  Week 4: Strongly disagree | 1 | 0
  Week 4: Disagree: number analyzed (Participants) | 11 | 18
  Week 4: Disagree | 0 | 0
  Week 4: Neither agree nor disagree: number analyzed (Participants) | 11 | 18
  Week 4: Neither agree nor disagree | 0 | 1
  Week 4: Agree: number analyzed (Participants) | 11 | 18
  Week 4: Agree | 6 | 8
  Week 4: Strongly agree: number analyzed (Participants) | 11 | 18
  Week 4: Strongly agree | 4 | 9
  Week 8: Strongly disagree: number analyzed (Participants) | 17 | 16
  Week 8: Strongly disagree | 0 | 0
  Week 8: Disagree: number analyzed (Participants) | 17 | 16
  Week 8: Disagree | 0 | 0
  Week 8: Neither agree nor disagree: number analyzed (Participants) | 17 | 16
  Week 8: Neither agree nor disagree | 0 | 1
  Week 8: Agree: number analyzed (Participants) | 17 | 16
  Week 8: Agree | 6 | 7
  Week 8: Strongly agree: number analyzed (Participants) | 17 | 16
  Week 8: Strongly agree | 11 | 8

9. Secondary Outcome: Percentage of Subjects Rating Each Device on Level of Convenience of Using the Device Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of convenience of using the device as "Extremely inconvenient", "Somewhat inconvenient", "Neutral/no opinion", "Somewhat convenient", or "Extremely convenient". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Extremely inconvenient | 0.0 | 2.0
  Week 4: Somewhat inconvenient | 8.7 | 18.0
  Week 4: Neutral/no opinion | 4.3 | 10.0
  Week 4: Somewhat convenient | 26.1 | 44.0
  Week 4: Extremely convenient | 60.9 | 26.0
  Week 8: Extremely inconvenient | 2.2 | 4.0
  Week 8: Somewhat inconvenient | 15.2 | 8.0
  Week 8: Neutral/no opinion | 8.7 | 8.0
  Week 8: Somewhat convenient | 39.1 | 34.0
  Week 8: Extremely convenient | 34.8 | 46.0

10. Secondary Outcome: Percentage of Subjects Rating Each Device on Level of Convenience of Storing the Device Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess how convenient it was to store the injection device. Subjects responded as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree" that the device was convenient to store.
Time Frame: Weeks 4 and 8
Population: FAS included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment. Here "Number of Participants Analyzed" signifies subjects evaluable for this outcome. Here results are presented by device sequence.
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 0.0 | 0.0
  Week 4: Disagree | 19.6 | 0.0
  Week 4: Neither agree nor disagree | 15.2 | 8.0
  Week 4: Agree | 34.8 | 58.0
  Week 4: Strongly agree | 30.4 | 34.0
  Week 8: Strongly disagree | 0.0 | 2.0
  Week 8: Disagree | 2.2 | 24.0
  Week 8: Neither agree nor disagree | 4.3 | 12.0
  Week 8: Agree | 54.3 | 40.0
  Week 8: Strongly agree | 39.1 | 22.0

11. Secondary Outcome: Percentage of Subjects Rating Each Device on Minimization of Safety Hazards Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess whether the device features help minimize safety hazards. Subjects responded as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 0.0 | 4.0
  Week 4: Disagree | 0.0 | 6.0
  Week 4: Neither agree nor disagree | 30.4 | 22.0
  Week 4: Agree | 34.8 | 48.0
  Week 4: Strongly agree | 34.8 | 20.0
  Week 8: Strongly disagree | 0.0 | 4.0
  Week 8: Disagree | 15.2 | 8.0
  Week 8: Neither agree nor disagree | 17.4 | 24.0
  Week 8: Agree | 39.1 | 32.0
  Week 8: Strongly agree | 28.3 | 32.0

12. Secondary Outcome: Percentage of Subjects Rating Each Device on Amount of Needle Anxiety While Using the Device Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their level of anxiety while giving themselves an injection with device. Subjects assessed their anxiety as "Not at all anxious", "A little anxious", "Moderately anxious", "Very anxious", "Extremely anxious". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Not at all anxious | 54.3 | 58.0
  Week 4: A little anxious | 19.6 | 26.0
  Week 4: Moderately anxious | 13.0 | 14.0
  Week 4: Very anxious | 6.5 | 2.0
  Week 4: Extremely anxious | 6.5 | 0.0
  Week 8: Not at all anxious | 47.8 | 44.0
  Week 8: A little anxious | 30.4 | 34.0
  Week 8: Moderately anxious | 8.7 | 12.0
  Week 8: Very anxious | 4.3 | 10.0
  Week 8: Extremely anxious | 8.7 | 0.0

13. Secondary Outcome: Percentage of Subjects Rating Each Device on Level of Satisfaction With Information Provided by the Trainer Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess whether the trainer provided easily understandable, unbiased and practical information about proper injection. Subjects responded as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 0.0 | 0.0
  Week 4: Disagree | 0.0 | 0.0
  Week 4: Neither agree nor disagree | 0.0 | 2.0
  Week 4: Agree | 32.6 | 38.0
  Week 4: Strongly agree | 67.4 | 60.0
  Week 8: Strongly disagree | 0.0 | 0.0
  Week 8: Disagree | 0.0 | 0.0
  Week 8: Neither agree nor disagree | 2.2 | 2.0
  Week 8: Agree | 19.6 | 28.0
  Week 8: Strongly agree | 78.3 | 70.0

14. Secondary Outcome: Percentage of Subjects Rating Each Device on Likelihood of Recommending the Device to Others Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked they would recommend injection device to others needing REBIF therapy. Subjects responded as "Very unlikely", "Unlikely", "Neutral/no opinion", "Likely", "Very likely". Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Very unlikely | 2.2 | 0.0
  Week 4: Unlikely | 10.9 | 8.0
  Week 4: Neutral/no opinion | 15.2 | 10.0
  Week 4: Likely | 23.9 | 42.0
  Week 4: Very likely | 47.8 | 40.0
  Week 8: Very unlikely | 4.3 | 10.0
  Week 8: Unlikely | 8.7 | 20.0
  Week 8: Neutral/no opinion | 13.0 | 8.0
  Week 8: Likely | 28.3 | 18.0
  Week 8: Very likely | 45.7 | 44.0

15. Secondary Outcome: Percentage of Subjects Rating Each Device on Overall Satisfaction With the Injection Device Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their overall satisfaction with using the device. Subjects responded as "Strongly disagree", "Disagree", "Neither agree nor disagree", "Agree", "Strongly agree" that they were satisfied with the device. Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: Strongly disagree | 2.2 | 2.0
  Week 4: Disagree | 15.2 | 6.0
  Week 4: Neither agree nor disagree | 10.9 | 8.0
  Week 4: Agree | 34.8 | 54.0
  Week 4: Strongly agree | 37.0 | 30.0
  Week 8: Strongly disagree | 2.2 | 8.0
  Week 8: Disagree | 4.3 | 16.0
  Week 8: Neither agree nor disagree | 10.9 | 16.0
  Week 8: Agree | 43.5 | 20.0
  Week 8: Strongly agree | 39.1 | 40.0

16. Secondary Outcome: Percentage of Subjects Rating Each Device on Ease of Use Based on User Trial Questionnaire (UTQ)
Description: The UTQ is a tool used to assess the ease-of-use of a device by the subject. Subjects were asked to assess their overall experience with using the device as "very difficult", "difficult", "neither easy nor difficult", "easy", or "very easy". Percentage of subjects who rated the overall use of device as very difficult", "difficult" or "neither easy nor difficult" were reported. Here results are presented by device sequence.
Time Frame: Weeks 4 and 8
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
percentage of subjects
  Week 4: very difficult | 0.0 | 0.0
  Week 4: difficult | 2.2 | 6.0
  Week 4: neither easy nor difficult | 23.9 | 14.0
  Week 8: very difficult | 2.2 | 4.0
  Week 8: difficult | 6.5 | 14.0
  Week 8: neither easy nor difficult | 15.2 | 18.0

17. Secondary Outcome: Change From Baseline in Multiple Sclerosis International Quality of Life (MusiQoL) Scores to Week 8
Description: The MusiQoL is a validated 31-item questionnaire describing 9 dimensions named according to its constitutive items:activities of daily living (8 items);psychological well-being (4 items);symptoms (3 items);friends relationships (4 items);family relationships (3 items);satisfaction with health care (RHCS 3 items);sentimental and sexual life (2 items);coping (2 items);and rejection (2 items). Each of the questions was answered using a 6-point Likert scale, defined as 1-Never/Not at all, 2-Rarely/A little, 3-Sometimes/Somewhat, 4-Often/A lot, 5-Always/Very much and 6-Not applicable. The scores of each dimension were obtained by computing mean of the item scores of dimension with negatively worded item scores reversed so that higher scores indicated higher health-related QoL. All 9 dimension scores were linearly transformed to a 0-100 scale,where higher score=higher health-related QoL. Global index score was computed as mean of the 9 dimension scores (range 0-100;higher score=higher QoL).
Time Frame: Baseline, up to Week 8
Population: FAS included all relapsing remitting multiple sclerosis subjects who received at least 1 injection of Rebif using either Rebif Rebidose or Rebiject II and had at least 1 post-baseline evaluation/assessment. Here "Number of Participants Analyzed" = subjects evaluable for this outcome, "Number Analyzed" = subjects evaluable for specified dimensions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | First Rebif Rebidose, Then Rebiject II | First Rebiject II, Then Rebif Rebidose
Number analyzed (Participants) | 46 | 50
score on a scale
  Baseline:Activities of daily living(ADL) | 69.0 (23.08) | 61.6 (26.64)
  Baseline:Psychological well-being (PWB) | 71.1 (24.38) | 68.2 (25.20)
  Baseline:Symptoms (SPT) | 71.3 (21.27) | 66.1 (22.84)
  Baseline:Friends relationships (RFr): number analyzed (Participants) | 41 | 46
  Baseline:Friends relationships (RFr) | 66.3 (19.00) | 64.9 (23.83)
  Baseline:Family relationships (RFa): number analyzed (Participants) | 45 | 49
  Baseline:Family relationships (RFa) | 81.3 (19.39) | 74.7 (21.85)
  Baseline: RHCS: number analyzed (Participants) | 42 | 45
  Baseline: RHCS | 63.7 (29.84) | 58.9 (34.50)
  Baseline:Sentimental and sexual life(SSL): number analyzed (Participants) | 46 | 48
  Baseline:Sentimental and sexual life(SSL) | 79.3 (24.75) | 74.0 (26.28)
  Baseline: Coping (COP): number analyzed (Participants) | 43 | 44
  Baseline: Coping (COP) | 93.6 (15.76) | 94.3 (10.60)
  Baseline: Rejection (REJ): number analyzed (Participants) | 45 | 49
  Baseline: Rejection (REJ) | 87.4 (21.37) | 88.8 (14.08)
  Baseline: Global index score: number analyzed (Participants) | 35 | 38
  Baseline: Global index score | 75.3 (14.52) | 72.8 (14.94)
  Change to Week 8: ADL: number analyzed (Participants) | 46 | 49
  Change to Week 8: ADL | 2.05 (13.773) | 4.51 (12.457)
  Change to Week 8: PWB: number analyzed (Participants) | 46 | 49
  Change to Week 8: PWB | 2.17 (13.124) | 2.98 (15.832)
  Change to Week 8: SPT: number analyzed (Participants) | 46 | 49
  Change to Week 8: SPT | 2.99 (12.271) | 3.61 (15.320)
  Change to Week 8: RFr: number analyzed (Participants) | 41 | 43
  Change to Week 8: RFr | -1.02 (21.746) | 0.68 (23.287)
  Change to Week 8: RFa: number analyzed (Participants) | 45 | 46
  Change to Week 8: RFa | -3.15 (13.211) | -2.54 (22.213)
  Change to Week 8: RHCS: number analyzed (Participants) | 39 | 37
  Change to Week 8: RHCS | 1.28 (21.228) | -4.39 (25.552)
  Change to Week 8: SSL: number analyzed (Participants) | 46 | 46
  Change to Week 8: SSL | 2.17 (9.612) | 3.26 (12.482)
  Change to Week 8: COP: number analyzed (Participants) | 41 | 42
  Change to Week 8: COP | 0.30 (10.639) | -0.30 (10.865)
  Change to Week 8: REJ: number analyzed (Participants) | 44 | 48
  Change to Week 8: REJ | 0.28 (19.737) | -0.52 (12.563)
  Change to Week 8: Global index score: number analyzed (Participants) | 32 | 26
  Change to Week 8: Global index score | 0.62 (7.275) | 0.87 (8.204)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 8
Arm/Group | Rebif Rebidose | Rebiject II
Serious Adverse Events (participants affected / at risk) | 1/95 | 0/97
Other Adverse Events (participants affected / at risk) | 3/95 | 5/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif Rebidose (N=95) | Rebiject II (N=97)
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif Rebidose (N=95) | Rebiject II (N=97)
Bruising at injection site-Left thigh (General disorders) | 0 | 1
Dosing error (General disorders) | 0 | 1
Numbness of right hand (General disorders) | 1 | 0
Redness (General disorders) | 0 | 1
Worsening of bunion (General disorders) | 0 | 1
Post bunionectomy pain (General disorders) | 0 | 1
Allergic reaction to artificial sweetener (aspartame) (General disorders) | 1 | 0
Tendonitis Right ring finger/hand (General disorders) | 0 | 1
Bilateral feet pain (General disorders) | 1 | 0
Right abdomen wall injection site reaction (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish or present any results from the Study to any third parties until i- EMD Serono publishes results from all sites participating in such Study;ii- Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned;or iii- twenty-four months following completion of the multi-site study at all sites, whichever comes first. Prior to publishing or presenting results from the study, PI must provide proposed publication to EMD Serono.